CLINICAL TRIAL: NCT02064218
Title: Evaluation of Some Emerging Biomarkers of Cardiovascular Risk Stratification in Hypertensive Patients: a 5-years Follow-up
Brief Title: Emerging Biomarkers in Hypertension
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Pavia (Other)
Collaborators: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Giuseppe Derosa, MD, PhD, University of Pavia
Other Study IDs: 20070002649
Record Dates: First submitted 2014-02-11; First posted 2014-02-17 (Estimated); Last update posted 2014-02-17 (Estimated); Status verified 2007-11

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Antihypertensive Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Hypertensive patients: Hypertensive patients naive to hypertensive treatment
  Interventions: Drug: Anti-hypertensive drugs
- healthy subjects: healthy subjects

INTERVENTIONS:
Drug: Anti-hypertensive drugs
  Groups: Hypertensive patients

SUMMARY:
First of all to evaluate the relationship between non-conventional biomarkers and essential hypertension; then to evaluate the effects of various anti-hypertensive drugs on blood pressure control and non-conventional biomarkers in naive hypertensive patients

ELIGIBILITY:
Inclusion Criteria:

* essential hypertension
* naive to treatment
* < 65 years

Exclusion Criteria:

* secondary hypertension
* previous cardiovascular events

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with naive essential hypertension aged < 65 years without previous cardiovascular events
Sampling Method: Probability Sample
Dates: Start 2007-11; Primary Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Blood pressure reduction | 5 years
  * Systolic Blood Pressure (SBP)
  * Diastolic Blood Pressure (DBP)

SECONDARY OUTCOMES:
Cardiovascular and metabolic biomarkers | 5 years
  * Lipoprotein (a) (Lp(a))
  * sRAGE (soluble Receptor for Advanced Glycation End-products)
  * sCD40L (soluble ligand of CD40)
  * MPO (myeloperoxidase)

OTHER OUTCOMES:
Evaluation of vascular stiffness | 5 years
  - Aortic Pulse Wave velocity (PWV)

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Derosa, MD, PhD, Principal Investigator — University of Pavia
Locations (1):
- IRCCS Policlinico S.Matteo Foundation, Pavia, Italy

REFERENCES:
- [Derived] Derosa G, Mugellini A, Pesce RM, D'Angelo A, Maffioli P. Barnidipine compared to lercanidipine in addition to losartan on endothelial damage and oxidative stress parameters in patients with hypertension and type 2 diabetes mellitus. BMC Cardiovasc Disord. 2016 Apr 12;16:66. doi: 10.1186/s12872-016-0237-z. PMID 27068332
- [Derived] Derosa G, Mugellini A, Pesce RM, D'Angelo A, Maffioli P. Perindopril and barnidipine alone or combined with simvastatin on hepatic steatosis and inflammatory parameters in hypertensive patients. Eur J Pharmacol. 2015 Nov 5;766:31-6. doi: 10.1016/j.ejphar.2015.09.030. Epub 2015 Sep 25. PMID 26407654
- [Derived] Derosa G, Mugellini A, Querci F, Franzetti I, Pesce RM, D'Angelo A, Maffioli P. Barnidipine or Lercanidipine on Echocardiographic Parameters in Hypertensive, Type 2 Diabetics with Left Ventricular Hypertrophy: A Randomized Clinical Trial. Sci Rep. 2015 Aug 5;5:12603. doi: 10.1038/srep12603. PMID 26243165
- [Derived] Derosa G, Mugellini A, Pesce RM, D'Angelo A, Maffioli P. A study about the relevance of adding acetylsalicylic acid in primary prevention in subjects with type 2 diabetes mellitus: effects on some new emerging biomarkers of cardiovascular risk. Cardiovasc Diabetol. 2015 Jul 30;14:95. doi: 10.1186/s12933-015-0254-8. PMID 26223257
- [Derived] Derosa G, Romano D, Bianchi L, D'Angelo A, Maffioli P. The effects of canrenone on inflammatory markers in patients with metabolic syndrome. Ann Med. 2015 Feb;47(1):47-52. doi: 10.3109/07853890.2014.969303. Epub 2014 Oct 16. PMID 25319120